CLINICAL TRIAL: NCT00881114
Title: A Prospective Phase II Clinical Trial to Use Pharmacogenetics (PGx) to Select Erbitux or Cisplatin to Treat Head and Neck Cancer
Brief Title: Study Using Pharmacogenetics to Select Treatment for Head and Neck Cancer
Acronym: PGx-SELECT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decided it was not feasible to conduct this study
Sponsor: Georgetown University (Other)
Responsible Party: John Deeken, MD, Georgetown University Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGx-SELECT; 2008-526
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2009-04

CONDITIONS: Head and Neck Cancer
Keywords: Head and neck cancer; pharmacogenetics; chemoradiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab (Experimental): patients with 2 or fewer genetic variants will receive cetuximab
  Interventions: Drug: Cetuximab
- Cisplatin (Experimental): Subjects with 3 to 8 genetic variants will receive cisplatin
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Intensity modulated radiation therapy with concurrent chemotherapy. Cisplatin will be administered at a dose of 100 mg/m2 during weeks 1, 4, and 7 of radiation therapy. Post treatment neck dissection will be performed if clinically indicated.
  Other Names: cis-diamminedichloridoplatinum(II); CDDP
  Arms: Cisplatin
Drug: Cetuximab — Intensity modulated Radiation Therapy with concurrent chemotherapy. Cetuximab will be administered beginning at a dose of 400 mg/m2 the week before radiation commences, then at a dose of 250 mg/m2 weekly during weeks 1 to 7. Post treatment neck dissection will be performed if clinically indicated.
  Other Names: Erbitux
  Arms: Cetuximab

SUMMARY:
This is a study for patients with head and neck cancer who will be receiving chemotherapy and radiation therapy for their disease. The purpose of this study is to see if the investigators can use genetic differences between patients to select the right drug to use with radiation therapy. This type of genetic testing is called pharmacogenetics.

Currently there are two drugs used to treat head and neck cancer that have provided a benefit when given with radiation compared to radiation alone in previous studies. These two drugs are cisplatin and cetuximab (Erbitux).

In this trial, the investigators will test whether genetic differences between patients can be used to pick which drug they should receive. A recent study that looked back to see how well patients with head and neck cancer responded to treatment with cisplatin showed that genetic differences in a few genes were associated with who did and who did not survive their cancer. The investigators are taking that finding and using it to test patients for these genetic differences to determine whether they should receive cisplatin or cetuximab. In other words, the investigators are trying to take what is essentially a flip of the coin choice between these two drugs, and instead use individual patient's genetic differences to make-and hopefully improve- this choice.

DETAILED DESCRIPTION:
Treatment-naive patients with locally advanced, non-metastatic (Stage III to IVB) squamous cell carcinoma of the head and neck who are candidates for concurrent chemoradiotherapy as primary therapy with curative intent will be enrolled. Patients will be genotyped for variations at four SNP loci in 3 genes involved in DNA nucleotide excision repair (ERCC1, ERCC2, and XRCC1). Patients with 3 to 8 variants will receive cisplatin, while patients with 2 or fewer variants will receive cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven squamous cell carcinoma of the head and neck, including of the oral cavity, oropharynx, hypopharynx, or larynx
* Locally advanced, Stage III or IVB disease and a candidate for primary therapy using chemotherapy and radiation with curative intent
* Patients with a diagnosis of 'unknown primary' will be eligible if chemoradiotherapy is primary modality of treatment
* No previous chemotherapy, radiation, or surgery for the diagnosis of head and neck cancer
* ECOG performance status 0 or 1
* Negative pregnancy test
* Hemoglobin >/= 8.0
* Absolute neutrophil count >/= 1500
* Platelet count >/= 100,000
* GFR > 50 mL/min
* Total bilirubin </= 1.5 upper limits of normal
* AST and ALT </= 2.5 times upper limits of normal
* No other current malignancy, other than basal cell skin cancer, squamous cell skin cancer, in situ cervical cancer, ductal or lobular in situ of the breast.
* Ability and willingness to give consent
* Subjects must in the opinion of the Investigator be capable of complying with the protocol

Exclusion Criteria:

* Primary tumors of the nasopharynx, sinuses, and salivary glands
* Acute treatment for an infection or other serious medical illness within 14 days prior to study entry
* Major surgery within 3 weeks prior to study entry
* Known hypersensitivity to cisplatin or cetuximab
* Patients who have any severe or uncontrolled medical conditions or other conditions that could affect their participation in this study including: unstable angina, serious uncontrolled cardiac arrhythmia, active or uncontrolled infectious disorder, myocardial infarction </= 6 months prior to study entry
* Psychiatric illness that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 36months

SECONDARY OUTCOMES:
Objective response | 36 months
Overall survival | 36 months
Toxicity | 8 weeks
Quality of Life | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: John Deeken, MD, Principal Investigator — Georgetown University